CLINICAL TRIAL: NCT06754930
Title: A Multicenter, Open Phase IB/II Clinical Study of Safety, Tolerability, and Efficacy of SHR-1826 in Combination With Other Anti-cancer Treatment in Patients With Non-small Cell Lung Cancer
Brief Title: A Study of SHR-1826 for Injection in Combination With Other Antitumor Therapies in Subjects With NSCLC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1826-201-LC
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Drug: SHR-1826; Drug: SHR-1316; Drug: SHR-9839; Drug: SHR-8068; Drug: Ametinib mesylate; Drug: BP-102; Drug: Carboplatin

INTERVENTIONS:
Drug: SHR-1826 — SHR-1826 for injection.
Drug: SHR-1316 — SHR-1316 for injection.
Drug: SHR-9839 — SHR-9839 for injection.
Drug: SHR-8068 — SHR-8068 for injection.
Drug: Ametinib mesylate — Ametinib mesylate.
Drug: BP-102 — BP-102 for injection.
Drug: Carboplatin — Carboplatin for injection.

SUMMARY:
This is an open label, multi-center, multiple dose Phase IB/II study to evaluate the safety, tolerability and efficacy of SHR-1826 for injection in subjects with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent.
2. 18-75 years older, no gender limitation.
3. Eastern Cooperative Oncology Group (ECOG) score: 0-1.
4. With a life expectancy ≥ 3 months.
5. Pathologically diagnosed NSCLC.
6. Be able to provide fresh or archived tumour tissue.
7. At least one measurable lesion according to RECIST v1.1.
8. Adequate organ function.
9. Contraception is required during clinical trials, and pregnancy tests must be negative for women of childbearing age within 7 days before the first dose.

Exclusion Criteria:

1. Meningeal metastasis history or clinical symptoms of central nervous system metastasis.
2. Previous or co-existing malignancies.
3. Spinal cord compression that was not treated radically by surgery and/or radiotherapy was excluded.
4. Uncontrollable tumor-related pain.
5. Have undergone major surgery other than diagnosis or biopsy within 28 days prior to the initial dosing; Minor traumatic surgery within 7 days prior to the first dosing.
6. Received other investigational drugs treatments 4 weeks prior to the initiation of the study treatment.
7. Unresolved CTCAE 5.0>grade 2 toxicities from previous anticancer therapy.
8. With poorly controlled or severe cardiovascular disease.
9. Active hepatitis B and hepatitis C.
10. Patients with a history of immunodeficiency.
11. Severe infection 30 days before the first dose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) | Screening up to study completion, an average of 1 year.
Adverse events (AEs) | Screening up to study completion, an average of 1 year.
Objective response rate (ORR) | Screening up to study completion, an average of 1 year.

SECONDARY OUTCOMES:
Disease control rate (DCR) | Screening up to study completion, an average of 1 year.
Duration of response (DoR) | Screening up to study completion, an average of 1 year.
Progression-free survival (PFS) | Screening up to study completion, an average of 1 year.
Overall survival (OS) | Screening up to study completion, an average of 1 year.
Drug resistant antibody (ADA) to SHR-1826 | Screening up to study completion, an average of 1 year.
Blood concentration of SHR-1826 | Screening up to study completion, an average of 1 year.
Blood concentration of free toxin | Screening up to study completion, an average of 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided